CLINICAL TRIAL: NCT03053505
Title: Two-arm, Interventional, Prospective, Open-label, Multi-center Trial to Evaluate the Safety & Effectiveness of FMT for Treatment of Adult Patients With Primary or Recurrent CDI, Using a Novel, Standardized Microbiota Transplantation System
Brief Title: A Novel Faecal Microbiota Transplantation System for Treatment of Primary and Recurrent Clostridium Difficile Infection
Acronym: FMTREAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sejtterapia Kozpont Kft. (Industry)
Collaborators: University of Debrecen (Other); Kenézy Gyula Korhaz es Rendelointezet (Unknown); Szabolcs-Szatmar-Bereg Megyei Korhaz es Egyetemi Oktatokorhaz (Unknown); Miskolci Semmelweis Korhaz es Egyetemi Oktatokorhaz (Unknown); Bacs-Kiskun Megyei Korhaz (Unknown); UD-Genomed Kft. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMT01
Record Dates: First submitted 2017-01-18; First posted 2017-02-15 (Actual); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Clostridium Difficile Infection
Keywords: fecal microbiota transplantation (FMT); Clostridium difficile infection; gut flora; human microbiome; colitis
MeSH Terms: conditions — Clostridium Infections; Colitis | interventions — Vancomycin; Fidaxomicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Recurrent CDI FMT (Experimental): Non-randomized group ("R") for treatment of recurrent CDI with FMT
  Interventions: Biological: faecal human microbiota transplant (FMT)
- Primary CDI antibiotic (Active Comparator): Randomized group ("F" AB) for the treatment of primary CDI with antibiotics (vancomycin or fidaxomicin)
  Interventions: Drug: Vancomycin or Fidaxomicin
- Primary CDI FMT (Experimental): Randomized group ("F" FMT) for the treatment of primary CDI with FMT
  Interventions: Biological: faecal human microbiota transplant (FMT)

INTERVENTIONS:
Biological: faecal human microbiota transplant (FMT) — Non-randomized group "R": Patients with recurrent CD infection are treated with FMT in this group.
  Randomized group "F"FMT: patients with initial CD infection who have severe disease or who are at high risk of recurrence or high risk of developing severe disease are treated with FMT.
  Other Names: FMT
  Arms: Primary CDI FMT; Recurrent CDI FMT
Drug: Vancomycin or Fidaxomicin — Randomized group "F"AB: patients with initial CD infection who have severe disease or who are at high risk of recurrence or high risk of developing severe disease are treated with antibiotics (vancomycin per os 125mg four times a day for 10 days) in this group. In case of treatment failure changes in antibiotic regime (e.g. fidaxomicin per os 200mg per two times a day for 10 days) will be allowed in the line with the recommendations of current CDI treatment guidelines(13).
  Arms: Primary CDI antibiotic

SUMMARY:
This study is a two-arm, interventional, prospective, open-label, multi-center clinical trial with randomized and non-randomized study groups to evaluate the safety and effectiveness of faecal microbiota transplantation (FMT) for the treatment of adult patients suffering from primary or recurrent Clostridium difficile infection (CDI), using a novel, standardized microbiota transplantation system.

DETAILED DESCRIPTION:
Clostridium difficile is an anaerobe, spore-forming bacillus. Infections with its toxin-producing strains are capable of causing CD associated enteral disease ranging in severity from mild diarrhea to fatal fulminant colitis. CD infection(CDI) occurs among patients who have taken antibiotics previously, suggesting that the normal gut flora is capable of preventing CDI. The disease is mainly treated with antibiotics, however, these antibiotics show high therapeutic failure and recurrence rates. There is significant interest in the development of alternative therapeutic strategies. Among the alternative methods only faecal microbiota transplantation (FMT) is gaining acceptance due to its excellent cure rate and low recurrence rate. FMT is a new approach to treating CDI, since no further antibiotics are administered, instead the normal gut flora being restored by administering faecal homogenisate from a healthy donor. Immediate risks of FMT are minimal, its efficacy is excellent,but further data is required about its short and long term safety, its most appropriate timing during the course of CDI and the optimal technical protocol for preparing the fecal homogenisate. In addition, the procedure is also challenging and the intervention itself is unappealing in nature. To address the challenges described above a novel faecal transplantation system has been designed (Burgin-Matic System, BMS), which is suitable for the production of faecal bacterial suspension in a standardized and controlled environment. Using this new approach, a multi-center,prospective,interventional clinical study involving two groups of patients has been designed: 1. In a non-randomized group("R") the safety and efficacy of FMT with the new, automated transplantation system will be assessed on 50 patients suffering from "R"ecurrent CDI. 2. In a randomized group ("F") FMT will be compared with the gold standard vancomycin treatment for 2x50 patients, with their "F"irst episode of CDI, suffering from severe infection or at risk of developing recurrent or severe disease and not responding to at least 72 hours of antibiotic treatment. In the non-randomized group("R"), the safety and efficacy of FMT will be assessed,with the hypothesis that FMT with the BMS is equally safe and effective(non-inferior)as reported in the international studies. In the randomized group ("F") primary endpoints will be the clinical cure rate at various time points, global cure rate at 10 weeks, time to clinical cure and time to global cure, while as secondary endpoints the cost effectiveness, quality of life, mortality will be assessed also. Our hypothesis is, that FMT with the BMS is superior to vancomycin treatment in terms of primary and secondary endpoints for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Group "R":- recurrent CDI;- positive stool toxin test within 72 hours before enrolment
* Group "F":- first (initial) episode of CDI;- enrolled patient falls in at least one of the following categories:high risk of recurrence or high risk of developing severe CDI or severe or life-threatening CDI;- patient requires hospitalization or CDI occurs during a hospital stay;- persisting symptoms despite least 72 hours of adequate antibiotic treatment;-positive stool CD toxin test obtained within 72 hours before screening;- in all cases, primary consideration must be given to the severity and pace of the patient's CDI when deciding whether early use of FMT is appropriate to prevent further clinical deterioration.

Exclusion Criteria:

* absence of either patient's or its legally authorized representative's informed consent
* inability or unwillingness to comply with protocol requirements
* severe co-morbidities, terminal underlying disease with a life expectancy of less than 90 days
* pregnancy or breastfeeding
* active gastroenteritis caused by microorganisms other than CD
* underlying chronic gastrointestinal disease that causes diarrhoea such as autonomic diabetic neuropathy, short bowel syndrome, faecal incontinence, active inflammatory bowel disease
* alimentary or over-the-counter drog allergy with previous anaphylactic reaction
* absolute contraindication to FMT

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Global cure rate at 10 weeks | 10 weeks after enrolment
Time to clinical cure | Through study completion, an average of 18 months
  The number of days between enrolment and the resolution of diarrhoea
Time to global cure | Through study completion, an average of 18 months
  The number of days between enrolment and the resolution of diarrhoea without relapse
Cure rate at 2 weeks | 2 weeks after enrolment
Cure rate at 4 weeks | 4 weeks after enrolment
Treatment failure rate | Through study completion, an average of 18 months
Recurrence rate 8 weeks after clinical cure | 8 weeks after clinical cure

SECONDARY OUTCOMES:
Number of adverse events (AE) | Through study completion, an average of 18 months
  Number of participants with treatment related adverse events
Number of serious adverse events (SAE) | Through study completion, an average of 18 months
  Number of participants with treatment related serious adverse events
Time of hospitalization | Through study completion, an average of 18 months
Days without diarrhoea during study period | Through study completion, an average of 18 months
Patient related quality of life | 0, 7, 14 days after enrolment
  Measured with EuroQoL 5Q-TL questionnaire
Professional acceptance | Through study completion, an average of 18 months
  A modified TSQM-14 questionnaire for assessing professional acceptance will be used during the study
General health survey for patients | 0, 7, 14 days after enrolment
  Measured with SF-36v2 questionnaire
Patient anxiety and depression | 0, 14, 70 days after enrolment
  Measured with HAD Scale (HADS)
Patient acceptance of treatment | 14,70 days after enrolment
  Measure with TSQM-14 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Gergely G Nagy, M.D., Ph.D., Study Chair — University of Debrecen; Zoltan Szilvassy, M.D., D.Sc., Study Director — University of Debrecen; Gyorgy Paragh, M.D., D.Sc., Principal Investigator — University of Debrecen; Istvan Varkonyi, M.D., Principal Investigator — Kenezy Gyula Korhaz es Rendelointezet; Zoltan Fulep, M.D., Principal Investigator — Bacs-Kiskun Megyei Korhaz; Laszlo Szegedi, M.D., Principal Investigator — Szabolcs-Szatmar-Bereg Megyei Korhaz es Egyetemi Oktatokorhaz; Tibor Pap, M.D., Principal Investigator — Miskolci Semmelweis Korhaz es Egyetemi Oktatokorhaz; Laszlo Nagy, M.D., D.Sc., Principal Investigator — UD-Genomed Kft.; Eva Rakoczi, M.D., Study Chair — Kenezy Gyula Korhaz es Rendelointezet; Judit Szabo, M.D., Ph.D., Study Chair — University of Debrecen; Maria Papp, M.D., Ph.D., Study Chair — University of Debrecen; Peter Vajo, Principal Investigator — Sejtterapia Kozpont Kft.
Locations (3):
- Hungary (3):
  - Miskolci Semmelweis Korhaz es Egyetemi Oktatokorhaz, Miskolc, B-a-z County
  - University of Debrecen, Clinical Centre, Debrecen, Hajdu-Bihar Megye
  - Szabolcs-Szatmar-Bereg Megyei Korhazak es Egyetemi Oktatokorhaz, Nyíregyháza, Szabocs-Szatmar-Bereg Megye

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Minkoff NZ, Aslam S, Medina M, Tanner-Smith EE, Zackular JP, Acra S, Nicholson MR, Imdad A. Fecal microbiota transplantation for the treatment of recurrent Clostridioides difficile (Clostridium difficile). Cochrane Database Syst Rev. 2023 Apr 25;4(4):CD013871. doi: 10.1002/14651858.CD013871.pub2. PMID 37096495